CLINICAL TRIAL: NCT03664674
Title: A Prospective, Randomized, Double Blind, Placebo-controlled, Multicenter, Phase 3 Efficacy and Safety Study of OTO-104 Given as a Single Intratympanic Injection in Subjects With Unilateral Meniere's Disease
Brief Title: Phase 3 Study of OTO-104 in Subjects With Unilateral Meniere's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otonomy, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 104-201811
Record Dates: First submitted 2018-08-31; First posted 2018-09-10 (Actual); Results first posted 2022-12-07 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-11

CONDITIONS: Meniere Disease
Keywords: Meniere's Disease; Vertigo; Endolymphatic Hydrops; Labyrinth Diseases; Ear Diseases; Otorhinolaryngologic Diseases
MeSH Terms: conditions — Meniere Disease; Vertigo; Endolymphatic Hydrops; Labyrinth Diseases; Ear Diseases; Otorhinolaryngologic Diseases

STUDY DESIGN:
Intervention Model Description: Randomized, Double-blind, Placebo-controlled, Multicenter
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- OTO-104 (Experimental)
  Interventions: Drug: OTO-104
- placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: OTO-104 — Single intratympanic injection of 12 mg dexamethasone
  Arms: OTO-104
Drug: Placebo — Single intratympanic injection of placebo
  Arms: placebo

SUMMARY:
The purpose of this study is to evaluate the effectiveness of OTO-104 for the treatment of Meniere's disease.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a diagnosis of unilateral Meniere's disease by 1995 American Academy of Otolaryngology - Head and Neck Surgery (AAOHNS) criteria and reports active vertigo for the 2 months prior to the study lead-in period.
* Subject has experienced active vertigo during the lead-in period.
* Subject has documented asymmetric sensorineural hearing loss.
* Subject agrees to maintain their current treatments for Meniere's disease while on-study.

Exclusion Criteria:

* Subject is pregnant or lactating.
* Subject has a history of immunodeficiency disease.
* Subject has a history of significant middle ear or inner ear surgery, or endolymphatic sac surgery in the affected ear.
* Subject has a history of tympanostomy tubes with evidence of perforation or lack of closure.
* Subject has a history of vestibular migraine.
* Subject has used an investigational drug or device in the 3 months prior to screening.
* Subject has previously been randomized to a clinical study of OTO-104.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2018-08-27 (Actual); Primary Completion 2020-12-22 (Actual); Study Completion 2020-12-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (65):
- United States (17):
  - Central California Clinical Research, Fresno, California
  - University of Colorado School of Medicine, Aurora, Colorado
  - Colorado ENT & Allergy, Colorado Springs, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - Ear, Nose and Throat Associates of South Florida, Boynton Beach, Florida
  - Ear Research Foundation, Sarasota, Florida
  - Tandem Clinical Research, Marrero, Louisiana
  - Michigan Ear Institute, Farmington Hills, Michigan
  - Saint Louis University, St Louis, Missouri
  - Dent Neurologic Institute, Amherst, New York
  - New York Eye and Ear Infirmary of Mount Sinai, New York, New York
  - Charlotte Eye Ear Nose & Throat Associates, P.A., Matthews, North Carolina
  - Piedmont Ear, Nose, and Throat Associates, PA, Winston-Salem, North Carolina
  - Medical University of South Carolina, Department of Otolaryngology, Charleston, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Intermountain Ear, Nose & Throat Specialists, Draper, Utah
  - West Virginia University School of Medicine, Morgantown, West Virginia
- Belgium (4):
  - Universitair Ziekenhuis Antwerpen - Ear-Nose-Throat Department, Edegem
  - UZ Gent - Ear-Nose-Throat Department, Ghent
  - UZ Leuven - Ear-Nose-Throat Department, Leuven
  - CHU de Liège - Ear-Nose-Throat Department, Liège
- Germany (11):
  - Uniklinik RWTH Aachen, Klinik für Hals-, Nasen-, Ohrenheilkunde und Plastische Kopf- und Halschirurgie, Aachen
  - Praxis Bad Essen, Bad Essen
  - Charité Universitätsmedizin Berlin, Berlin
  - HNO Zentrum am Kudamm, Berlin
  - HNO-Praxis Göttingen, Göttingen
  - HNO Praxis am Neckar, Heidelberg
  - HNO Praxis Dres. med. Florian Heimlich und Angelika Witzel-Heimlich, Heidelberg
  - Universitätsklinikum Mannheim, Mannheim
  - HNO Praxis Dr. med. Roger Fisher, Markkleeberg
  - Klinikum der Universität München, München
  - Universitätsklinikum Ulm, HNO-Klinik. Kopf-Hals-Chirurgie, Ulm
- Italy (4):
  - U.O. di Otorinolaringoiatria Universitaria, Bari, NAP
  - Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico - U.O.S.D. Audiologia, Milan
  - Unità Operativa di Otorinolaringoiatria, Piacenza
  - Azienda Ospedaliera-Universitaria Sant' Andrea; Dipartimento Organi di Senso-U.O.C. Otorinolaringoiatria, Roma
- Poland (7):
  - 10 Wojskowy Szpital Kliniczny z Polikliniką SP ZOZ Oddział, Bydgoszcz
  - Centrum Medyczne ZDROWA, Krakow
  - Centrum Medyczne PROMED, Krakow
  - MT Medic Specjalistyczna Praktyka Lekarska Tomasz Stapiński, Krosno
  - ETG Łódź, Lodz
  - Centrum Słuchu i Mowy Sp. z o.o., Nadarzyn
  - Kliniczny Szpital Wojewódzki Nr 1 im. Fryderyka Chopina, Rzeszów
- Spain (4):
  - Agencia Pública Empresarial Sanitaria Hospital de Poniente, El Ejido, Almería
  - Hospital Universitario de Getafe, Getafe, Madrid
  - Hospital Universitario Virgen de las Nieves, Granada
  - Hospital Universitario Virgen Macarena, Seville
- Turkey (Türkiye) (8):
  - Hacettepe Universitesi Tip Fakultesi Kulak Burun Bogaz Hastaliklari Anabilim Dali, Ankara
  - Baskent Universitesi Ankara Hastanesi, Kulak Burun Bogaz Hastaliklari Ana Bilim Dali, Ankara
  - Bayindir Hastanesi Sogutozu, Kulak Burun Bogaz Bas ve Boyun Cerrahisi Bolumu, Ankara
  - Uludag Universitesi Saglik Uygulama ve Arastirma Merkezi, Kulak Burum Bogaz Hastaliklari Ana Bilim Dali, Bursa
  - Istanbul Universitesi Istanbul Tip Fakultesi Kulak Burun Bogaz Hastaliklari Anabilim Dali, Istanbul
  - Acibadem Maslak Hastanesi Kulak Burun Bogaz Bolumu, Istanbul
  - Ege Universitesi Tip Fakultesi Kulak Burun Bogaz Hastaliklari Anabilim Dali, Izmir
  - Dokuz Eylul Universitesi Tip Fakultesi Tip Bilimleri Bolumu Kulak Burun Bogaz Anabilim Dali, Izmir
- United Kingdom (10):
  - Ninewells Hospital and Medical School, Dundee, Angus
  - Royal Victoria Hospital, Belfast
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - University Hospital of Wales, Cardiff
  - Gloucestershire Royal Hospital, Gloucester
  - University Hospitals of Leicester NHS Trust, Leicester Royal Infirmary, Leicester
  - Guy's and St Thomas' NHS Foundation Trust, London
  - Manchester Head and Neck Centre, Peter Mount Building, Manchester
  - Norfolk & Norwich University Hospital, Norwich
  - The Royal Hallamshire Hospital, Sheffield

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Phillips J, Mikulec AA, Robinson JM, Skarinsky D, Anderson JJ. Efficacy of Intratympanic OTO-104 for the Treatment of Meniere's Disease: The Outcome of Three Randomized, Double-Blind, Placebo-Controlled Studies. Otol Neurotol. 2023 Jul 1;44(6):584-592. doi: 10.1097/MAO.0000000000003886. Epub 2023 Apr 22. PMID 37185596

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 148 subjects were randomized and 148 subjects received study drug. The most common reason for screen failure was that there was not a sufficient number of definitive vertigo days in the 28-day lead-in period.
Pre-assignment Details: In addition to meeting all screening visit inclusion criteria, potential subjects had to experience and record at least 4 and a maximum of 22 definitive vertigo day (DVD) during the 4-week lead-in period, where no intervention was administered. Also, the subject needed to complete at least 22 of 28 diary entries during this lead-in period. A DVD was defined as each day the subject recorded a vertigo episode lasting at least 20 minutes corresponding to a vertigo score of 2 or more.
Period: Overall Study
Arm/Group | OTO-104 | Placebo
Started | 73 | 75
Completed | 70 | 73
Not Completed | 3 | 2
Not completed — Adverse Event | 1 | 1
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Population: This population is designated as the Safety Analysis Set, which is comprised of all subjects that were randomized and received study drug. They are grouped based on what they received, not what they were randomized to receive.
Groups:
- Total: Total of all reporting groups
Arm/Group | OTO-104 | Placebo | Total
Number analyzed (Participants) | 73 | 75 | 148
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 51 | 57 | 108
  >=65 years | 22 | 18 | 40
Age, Continuous [Median (Full Range); unit: years] | 57.0 [27 to 75] | 57.0 [26 to 83] | 57.0 [26 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 44 | 88
  Male | 29 | 31 | 60
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 71 | 73 | 144
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 73 | 71 | 144
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 3 | 3
Region of Enrollment [Number; unit: participants]
  Turkey | 3 | 8 | 11
  Belgium | 3 | 6 | 9
  United States | 8 | 13 | 21
  Poland | 31 | 29 | 60
  Italy | 7 | 5 | 12
  United Kingdom | 7 | 9 | 16
  Germany | 11 | 4 | 15
  Spain | 3 | 1 | 4
Duration of Meniere's disease [Count of Participants; unit: Participants]
  <5 years | 61 | 53 | 114
  6-10 years | 9 | 13 | 22
  11-15 years | 0 | 4 | 4
  >15 years | 3 | 5 | 8

OUTCOME MEASURES:

1. Primary Outcome: 28-Day Average DVD at Week 12 (Month 3)
Description: The count of definitive vertigo days for Week 12 was determined during the 4-week period between Weeks 9 and 12. The 28-day average DVD was derived for each subject and visit by summing each subject's number of DVD counts within the 4-week interval, dividing by the number of completed diary days, and multiplying by 28.
Time Frame: 3 months
Measure: Least Squares Mean (95% Confidence Interval); unit: DVD
Groups:
- OTO-104 Intent to Treat; Placebo Intent to Treat: Includes all randomized subjects who received study drug. Subjects were included in the treatment group to which they were randomized regardless of the actual study drug received.
Arm/Group | OTO-104 Intent to Treat | Placebo Intent to Treat
Number analyzed (Participants) | 73 | 75
DVD | 2.869 [2.109 to 3.903] | 3.577 [2.641 to 4.844]
Statistical Analysis 1: Comparison: OTO-104 Intent to Treat vs Placebo Intent to Treat; Test type: Superiority; p = 0.312, Regression, Linear — Generalized Linear Model - Negative Binomial Regression Model with count data by subject transformed using the log-link function; The parameter estimate + conf. int. results back-transform to the ratio of adjusted mean DVDs (OTO-104/Placebo) to be 0.802 (0.523, 1.230); Mean Difference (Net) = -0.221, 95% CI 2-sided [-0.648 to 0.207], Standard Error of Mean 0.218

2. Secondary Outcome: Impact of Vertigo Experience on Daily Activities at Week 12 (Month 3) - The Number of Days Sick at Home or Bedridden
Description: The count of days sick at home or bedridden for subsequent intervals was determined during the 4-week period between each visit. The count of days sick at home or bedridden was computed as the sum of the days in the Sick at home and Bedridden categories for each 4-week interval and was standardized to 28 days by multiplying by 28 days and dividing by the number of non-missing diary entries.
Time Frame: 3 Months
Measure: Mean (Standard Deviation); unit: days
Arm/Group | OTO-104 Intent to Treat | Placebo Intent to Treat
Number analyzed (Participants) | 73 | 75
days | 0.998 (2.1521) | 1.643 (2.5783)

3. Secondary Outcome: Otoscopic Examination - Presence of Perforation in the Treated Ear at Week 12 (Month 3) Final Visit
Description: Ear examinations were done at every visit. One of the important safety endpoints was an observation of a perforation in the ear drum did not heal properly after the injection. Reported here are the Week 12 (Month 3) final visit.
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | OTO-104 | Placebo
Number analyzed (Participants) | 73 | 75
Participants | 0 | 0

4. Secondary Outcome: Audiometry - Shift in Air-Bone Gap at 1000 Hz From Baseline to Week 12 (Month 3)
Description: The number of subjects with a change in air-bone gap from Baseline to Week 12 (Month 3) from no impairment at baseline (<= 10 dB) to impairment at Month 3 (>10 dB) when measured at 1000 Hz.
Time Frame: Week 12 (Month 3)
Population: Subjects that had no impairment at the Baseline visit (air-bone gap <= 10 dB)
Measure: Count of Participants; unit: Participants
Arm/Group | OTO-104 | Placebo
Number analyzed (Participants) | 55 | 58
Participants | 5 | 7

5. Secondary Outcome: Audiometry - Shift in Air-Bone Gap at 2000 Hz From Baseline to Week 12 (Month 3)
Description: The number of subjects with a change in air-bone gap from Baseline to Week 12 (Month 3) from no impairment at baseline (<= 10 dB) to impairment at Month 3 (>10 dB) when measured at 2000 Hz.
Time Frame: Week 12 (Month 3)
Population: Subjects that had no impairment at the Baseline visit (air-bone gap <= 10 dB)
Measure: Count of Participants; unit: Participants
Arm/Group | OTO-104 | Placebo
Number analyzed (Participants) | 62 | 64
Participants | 4 | 4

6. Secondary Outcome: Audiometry - Shift in Air-Bone Gap at 4000 Hz From Baseline to Week 12 (Month 3)
Description: The number of subjects with a change in air-bone gap from Baseline to Week 12 (Month 3) from no impairment at baseline (<= 10 dB) to impairment at Month 3 (>10 dB) when measured at 4000 Hz.
Time Frame: Week 12 (Month 3)
Population: Subjects that had no impairment at the Baseline visit (air-bone gap <= 10 dB)
Measure: Count of Participants; unit: Participants
Arm/Group | OTO-104 | Placebo
Number analyzed (Participants) | 50 | 53
Participants | 2 | 9

ADVERSE EVENTS:
Time Frame: Reported or observed during or after dosing with the study drug up until end of study (Week 12/Month 3).
Arm/Group | OTO-104 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/73 | 0/75
Serious Adverse Events (participants affected / at risk) | 2/73 | 2/75
Other Adverse Events (participants affected / at risk) | 26/73 | 27/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OTO-104 (N=73) | Placebo (N=75)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
Uterine Haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Meniere's disease (Ear and labyrinth disorders) | 0 (0) | 1 (1) — Subject was also hospitalized for hypertension the day after being discharged following recovery of exacerbation of Meniere's disease.
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OTO-104 (N=73) | Placebo (N=75)
Meniere's disease (Ear and labyrinth disorders) | 6 (6) | 6 (6)
Tinnitus (Ear and labyrinth disorders) | 5 (5) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 4 (4) | 7 (7)
Ear Discomfort (Ear and labyrinth disorders) | 2 (2) | 2 (2)
Ear Pain (Ear and labyrinth disorders) | 1 (1) | 4 (4)
Tympanic Membrane Disorders (Ear and labyrinth disorders) | 0 (0) | 2 (2)
Upper Respiratory Infection (Infections and infestations) | 2 (2) | 2 (2)
Nasopharyngitis (Infections and infestations) | 1 (1) | 2 (2)
Limb Injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-30): https://cdn.clinicaltrials.gov/large-docs/74/NCT03664674/Prot_SAP_000.pdf